CLINICAL TRIAL: NCT02944604
Title: The Efficacy and Safety of PEG-rhG-CSF（Pegylated Recombinant Human Granulocyte Colony Stimulating Factor)in Patients With Breast Cancer Who Were Treated With Intensive Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-20160314
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Breastcancer
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

ARMS (1):
- PEG-rhG-CSF (Experimental): Patients with breast cancer who were treated with intensive chemotherapy received PEG-rhG-CSF.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of PEG-rhG-CSF in patients with breast cancer who were treated with intensive chemotherapy for prevention of neutrophil reduction.

ELIGIBILITY:
Inclusion Criteria:

1.18-65 years old, gender no limited.

2.Breast cancer diagnosed by pathology.

3.Did not receive chemotherapy previously and plans to receive 4 cycles intensive EC (epirubicin, cyclophosphamide) treatment.

4.No obvious blood system disease, ANC(absolute neutrophil count)≥ 1.5 × 10^9/L, PLT（Platelet）≥80×10^9 /L, Hb（hemoglobin）≥75g/L, WBC（White blood cell ）≥3×109/L, and no bleeding tendency.

5.KPS (Karnofsky performance status) score≥70.

6.Expected survival≥3 months.

7.Written informed consent are acquired.

Exclusion Criteria:

1. Severe or uncontrolled infection.
2. Sensitive to the product or other genetically engineered biological products from Escherichia coli strains.
3. Mental or nervous system disorders.
4. Severe heart, lung and central nervous system disorders.
5. Pregnant or lactating women.
6. TBIL(total bilirubin ), ALT（alanine aminotransferase）,AST（glutamic-oxalacetic transaminase） > 2.5×ULN（upper limit of normal）; if it were caused by liver metastases, TBIL, ALT,AST >5×ULN.
7. Cr（creatinine） >1.5×ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of chemotherapy delay | 60 days after the first chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China